CLINICAL TRIAL: NCT01515800
Title: S1105, Randomized Trial Of Text-Messaging Intervention To Reduce Early Discontinuation Of Adjuvant Aromatase Inhibitor Therapy In Women With Early Stage Breast Cancer
Brief Title: S1105: Text-Messaging Intervention to Reduce Early Discontinuation of AI Therapy in Women With Early-Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CDR0000723653; S1105 (Other: SWOG); U10CA037429 (NIH)
Record Dates: First submitted 2012-01-21; First posted 2012-01-24 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Text message reminder (Experimental): Patients undergo a text message education checklist involving confirmation of cellular telephone capability to receive text messages, how to retrieve and read messages, including a confirmation evaluation, at baseline and at any time a patient obtains a new cellular telephone. Patients then receive a text message twice a week at 8 o'clock in the morning (for each time zone) for up to 3 years. Additionally, patients receive standard follow-up care.
  Interventions: Behavioral: Text message reminder
- No text message reminder (No Intervention): Patients receive standard follow-up care.

INTERVENTIONS:
Behavioral: Text message reminder — Receive text message
  Arms: Text message reminder

SUMMARY:
RATIONALE: Measuring how text-message affects treatment compliance in women with breast cancer may help doctors plan the best treatment.

PURPOSE: This randomized trial studies how well text-message works in reducing early discontinuation of aromatase inhibitor therapy in patients with early-stage breast cancer who underwent breast surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of a reminder message, sent by text message to mobile phones twice weekly, to improve adherence to adjuvant aromatase inhibitor (AI) therapy as determined by urinary AI levels in women with early-stage hormone-sensitive breast cancer versus usual care.

Secondary

* To compare the effect of a reminder message sent twice weekly to mobile phones as compared to usual care to improve adherence to adjuvant AI therapy according to self-report.
* To explore the efficacy of the text message intervention for reducing early discontinuation as compared to usual care at 12, 24, and 36 months of adjuvant AI therapy in subgroups of breast cancer patients as defined by age group, stage, year of therapy, education, race/ethnicity, teaching hospital versus community hospital, AI-related side effects (as determined by serial questionnaires), insurance status, and prescription co-pay status.
* To explore the reasons for early discontinuation of AI therapy in those who do discontinue in the intervention and control group by querying quality of life as assessed by the Functional Assessment of Cancer Therapy-Endocrine Subscales (FACT-ES) and symptoms and other issues related to hormonal therapy at each follow-up visit, using the Brief Pain Inventory (BPI-SF), and at annual visits the Beliefs about Medicine Questionnaire (BQM) and the Treatment Satisfaction Questionnaire for Medication (TSQM).
* To conduct a sensitivity analysis assessing time to last evidence of adherence.

OUTLINE: This is a multicenter study. Patients are stratified according to length of time on aromatase inhibitor (AI) (< 12 months vs 12-24 months), and type of AI (anastrozole vs letrozole vs exemestane). Patients are randomized to 1 of 2 intervention arms.

* Arm I: Patients undergo a text message education checklist involving confirmation of cellular telephone capability to receive text messages, how to retrieve and read messages, including a confirmation evaluation, at baseline and at any time a patient obtains a new cellular telephone. Patients then receive a text message twice a week at 8 o'clock in the morning (for each time zone) for up to 3 years.
* Arm II: Patients receive standard follow-up care. Patients undergo urine sample collection at baseline and periodically during study for aromatase inhibitor level analysis and future translational studies.

Patients complete the Functional Assessment of Cancer Therapy-Endocrine Subscales (FACT-ES), the Brief Pain Inventory (BPI-SF), Beliefs about Medicine Questionnaire (BQM), and the Treatment Satisfaction Questionnaire for Medication (TSQM) questionnaires at baseline and periodically during study. Patients in arm I also complete the Cell Phone and Text Messaging Use Questionnaire at baseline and periodically during study.

In both arms, patients are followed up every 3 months for up to 3 years from registration.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients must be women with a diagnosis of histologically confirmed, primary invasive, hormone-sensitive (estrogen receptor-positive [ER]/progesterone receptor [PR]-positive) adenocarcinoma of the breast (Stage I, II or III) with no evidence of recurrent or metastatic disease (M0)
* Patients must have a mobile phone that can receive text messages and must currently use or be willing to learn to use text messaging

PATIENT CHARACTERISTICS:

* Patients must be postmenopausal, as defined by at least one of the following:

  * ≥ 12 months since the last menstrual period
  * Prior bilateral oophorectomy
  * Previous hysterectomy with one or both ovaries left in place (or previous hysterectomy in which documentation of bilateral oophorectomy is unavailable) AND follicle-stimulating hormone (FSH) values consistent with the institutional normal values for the postmenopausal state; FSH levels must be obtained within 28 days prior to registration
* Patients must be willing to provide urine specimen to test for the presence of aromatase inhibitor within 28 days of randomization and at each 3-month clinic visit for 3 years
* Patients must have the ability to speak and read English
* Patients must have a Zubrod performance status of 0 - 2
* No other prior malignancy (i.e., other than as noted on disease characteristics) is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for > 5 years
* Patients are allowed to participate in another clinical trial as long as it does not interfere with daily intake of aromatase-inhibitor therapy

PRIOR CONCURRENT THERAPY:

* Patients must be post adjuvant chemotherapy (if to be utilized) and primary curative surgery and must have recovered from all side-effects of the surgery

  * Trastuzumab (Herceptin) given alone after cytotoxic chemotherapy is considered adjuvant chemotherapy; patients would be eligible upon completion of Herceptin as long as the other eligibility criteria are met
* Patients must be currently taking an aromatase inhibitor (AI), have completed at least one month of AI therapy, be within the first 5 years of planned AI therapy, and have at least 3 years remaining before completion of planned AI therapy

Exclusion criteria: Insufficient evidence of post-menopausal status; metastatic or recurrent disease; currently receiving chemotherapy.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2012-05; Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Time to first evidence of adherence failure (discontinuation) | Every 3 months after randomization

SECONDARY OUTCOMES:
Adherence effect of text message compared to usual care using the patient self-report responses to AI Usage form | Every 3 months after randomization
Relationship between randomized arm and various participant, site and health insurance characteristics | Every 3 months after randomization
  Relationship between randomized arm and the following factors: age group, stage, years of therapy, education, race/ethnicity, teaching hospital versus community hospital, AI-related side effects, insurance status, and prescription co-pay status.
Reasons for early discontinuation of AI therapy among intervention arm and control arm as assessed by quality-of-life questionnaires | Every 3 months after randomization
Time to last evidence of adherence | Every 3 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Alfred I. Neugut, MD, PhD, Principal Investigator — Herbert Irving Comprehensive Cancer Center
Locations (204):
- United States (204):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Kaiser Permanente - Fremont, Fremont, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Kaiser Permanente Fresno Medical Center, Fresno, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Oncare Hawaii, Incorporated - Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Highland Clinic, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Mercy Clinic Cancer and Hematology - Rolla, Rolla, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - Presbyterian Cancer Treatment Center at Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Falck Cancer Center at Arnot Ogden Medical Center, Elmira, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Winthrop University Hospital, Mineola, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Waverly Hematology Oncology, Cary, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Swedish Medical Center - Issaquah Campus, Issaquah, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming

REFERENCES:
- [Derived] Hershman DL, Unger JM, Hillyer GC, Moseley A, Arnold KB, Dakhil SR, Esparaz BT, Kuan MC, Graham ML 2nd, Lackowski DM, Edenfield WJ, Dayao ZR, Henry NL, Gralow JR, Ramsey SD, Neugut AI. Randomized Trial of Text Messaging to Reduce Early Discontinuation of Adjuvant Aromatase Inhibitor Therapy in Women With Early-Stage Breast Cancer: SWOG S1105. J Clin Oncol. 2020 Jul 1;38(19):2122-2129. doi: 10.1200/JCO.19.02699. Epub 2020 May 5. PMID 32369401